CLINICAL TRIAL: NCT02013206
Title: An Parallel Phase II Study of Tarceva (Erlotinib) in Patients With Advanced Non-small Cell Lung Cancer (Stage IIIB/IV) Not Pre-treated by Chemotherapy Including Dose Escalation to Toxicity in Current and Former Smokers
Brief Title: A Study of Tarceva (Erlotinib) in Patients With Advanced Non-Small Cell Lung Cancer Naive to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO18660
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Never Smokers (Experimental): Never Smokers (participants who smoked ≤ 100 cigarettes in entire lifetime or had never smoked cigarettes) received erlotinib [Tarceva] 150 mg orally daily until disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib [Tarceva]
- Current/Former Smokers (Experimental): Current Smokers (participants who smoked > 100 cigarettes in entire lifetime and either quit smoking < 1 year ago or were currently smoking) or Former Smokers (participants who smoked > 100 cigarettes in entire lifetime and quit smoking ≥ 1 year ago) received erlotinib [Tarceva] 150 mg orally daily, increasing to a maximum of 300 mg orally daily until disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: erlotinib [Tarceva] — Erlotinib tablets taken orally once daily in the morning.
  Other Names: Tarceva

SUMMARY:
This study will evaluate the efficacy and safety of Tarceva in two groups of patients with non-small cell lung cancer who have not been pre-treated with chemotherapy. One group, consisting of patients who have never smoked, will receive Tarceva 150 mg/day, and the other group, consisting of current/former smokers, will receive Tarceva 150 mg/day increasing to a maximum of 300 mg/day. The anticipated time on study treatment is 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* histologically documented advanced non-small cell lung cancer (stage IIIB/IV);
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* no previous chemotherapy.

Exclusion Criteria:

* previous therapy which acts on Epidermal Growth Factor Receptor (EGFR) axis;
* clinical evidence of brain metastasis;
* any unstable systemic disease;
* unable to take oral medication;
* any significant ophthalmological abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (10):
- France (2):
  - Marseille
  - Villejuif
- Hamburg, Germany
- Italy (2):
  - Milan
  - Rozzano
- Netherlands (2):
  - Amsterdam
  - Maastricht
- Spain (2):
  - Barcelona
  - Madrid
- Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Current/Former Smokers | Never Smokers
Started | 29 | 23
Received Study Drug | 26 | 23
Completed | 2 (3 Patients were on-going at clinical cut-off. Not Completed=patients who discontinued treatment.) | 1
Not Completed | 27 | 22
Not completed — Progressive disease (PD) | 14 | 17
Not completed — Symptomatic deterioration | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Patient refusal | 2 | 0
Not completed — Patient non-compliance | 1 | 0
Not completed — Death | 1 | 2
Not completed — Other reasons off treatment | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Current/Former Smokers | Never Smokers | Total
Number analyzed (Participants) | 29 | 23 | 52
Age, Continuous [Mean (Full Range); unit: years] | 64 [38 to 83] | 66 [42 to 88] | 65 [38 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 14 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Non-Progression Rate (NPR) at 8 Weeks
Description: Non-Progressive Rate (NPR) was defined as the percentage of participants without progression (had stable disease (SD) or better) based on (Response Evaluation Criteria in Solid Tumours (RECIST) criteria 8 weeks after start of treatment. Diagnosis of Progressive Disease (PD) was made by objective criteria (RECIST criteria) on the target lesion(s), or by documenting, with Computerised Tomography/Magnetic Resonance Imaging (CT/MRI) scans, the presence of newly occurring lesion(s) arising outside the scanned areas of the target lesions. PD required at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Week 8
Population: Intent-to-Treat Population included all registered participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Current/Former Smokers | Never Smokers
Number analyzed (Participants) | 29 | 23
percentage of participants | 41.4 [23.5 to 61.1] | 65.2 [42.7 to 83.6]

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants with Complete Response (CR) or Partial Response (PR) by Response Evaluation Criteria in Solid Tumours (RECIST). The best overall response was the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). The patient's best response assignment depended on the achievement of both measurement and confirmation criteria. To be assigned the status of PR or CR, changes in tumour measurements were to be confirmed by repeated assessments no less than 4 weeks after the criteria for response were first met.
  CR was defined as the disappearance of all target lesions; for non-target lesions disappearance of lesions and normal tumour marker levels. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, using as reference the Baseline sum LD.
Time Frame: Up to 2 years
Population: Intent-to-Treat Population included all registered participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Current/Former Smokers | Never Smokers
Number analyzed (Participants) | 29 | 23
percentage of participants | 17 [5.9 to 35.8] | 35 [16.4 to 57.3]

3. Secondary Outcome: Disease Control Rate
Description: Disease Control Rate was defined as the percentage of participants with Complete Response (CR), Partial Response (PR) or Stable Disease (SD) by Response Evaluation Criteria in Solid Tumours (RECIST). CR was defined as the disappearance of all target lesions; for non-target lesions disappearance of lesions and normal tumour marker levels. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, using as reference the Baseline sum LD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started; for non-target lesions persistence of one or more non-target lesion(s) and/or maintenance of tumour marker level above the normal limits.
Time Frame: Up to 2 years
Population: Intent-to-Treat Population included all registered participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Current/Former Smokers | Never Smokers
Number analyzed (Participants) | 29 | 23
percentage of participants | 41 [23.5 to 61.1] | 65 [42.7 to 83.6]

4. Secondary Outcome: Duration of Response
Description: Duration of overall response was defined as the time in months from Complete Response (CR) or Partial Response (PR) by Response Evaluation Criteria in Solid Tumours (RECIST) until the first date Progressive Disease (PD) was objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started) or until the date of death. CR was defined as the disappearance of all target lesions; for non-target lesions disappearance of lesions and normal tumour marker levels.PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, using as reference the Baseline sum LD. PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 2 years
Population: Participants from the Intent-to-Treat (ITT) Population, that included all participants, with CR or PR. Patients still responding to treatment at the time of analysis were treated as censored observations for duration of response on the date of the last tumour assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Current/Former Smokers | Never Smokers
Number analyzed (Participants) | 5 | 8
months | 13.1 [4.6 to 13.1] | 5.7 [4.0 to NA] — 95% Confidence Interval Upper limit was not estimated due to the small number of participants.

5. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from start of treatment until the first date criteria for Progressive Disease (PD) was met (taking as reference the smallest measurements recorded since the treatment started). Diagnosis of PD was made by objective criteria (RECIST criteria) on the target lesion(s), or by documenting, with Computerised Tomography/Magnetic Resonance Imaging (CT/MRI) scans, the presence of newly occurring lesion(s) arising outside the scanned areas of the target lesions. PD required at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 2 years
Population: Safety Population included all registered patients who received at least 1 dose of study treatment and had at least 1 safety follow-up. Patients without PD at the time of analysis were censored on the date of the last tumour assessment. Patients without PD who received a second anti-cancer therapy were censored prior to start of new therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Current/Former Smokers | Never Smokers
Number analyzed (Participants) | 26 | 23
months | 1.9 [1.0 to 5.6] | 5.5 [3.4 to 7.3]

6. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival (PFS) was defined as the time in months from the start of treatment until the first date criteria for Progressive Disease (PD) were met (taking as reference the smallest measurements recorded since the treatment started), or the date of death for any reason in the absence of PD. Diagnosis of PD was made by objective criteria (RECIST criteria) on the target lesion(s), or by documenting, with Computerised Tomography/Magnetic Resonance Imaging (CT/MRI) scans, the presence of newly occurring lesion(s) arising outside the scanned areas of the target lesions.
Time Frame: Up to 2 years
Population: Safety Population included all registered participants who received at least one study treatment and had at least one safety follow-up. Patients without PD at the time of analysis were censored on the date of the last tumour assessment. Patients without PD who received a second anti-cancer therapy were censored prior to start of new therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Current/Former Smokers | Never Smokers
Number analyzed (Participants) | 26 | 23
months | 1.9 [1.0 to 5.6] | 4.1 [3.4 to 5.7]

7. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months from the start of treatment to the date of death irrespective of the cause of death.
Time Frame: Up to 2 years
Population: Safety Population included all participants with at least one study treatment and had at least one safety follow-up. Patients who had not died at the time of the final analysis were censored at the date of last contact.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Current/Former Smokers | Never Smokers
Number analyzed (Participants) | 26 | 23
months | 9.9 [5.6 to 14.0] | 13.9 [8.9 to 18.0]

8. Secondary Outcome: Safety: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events. A SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: Up to 2 years
Population: Safety Population included all registered participant who received at least one study treatment and had at least one safety follow-up.
Measure: Number; unit: participants
Arm/Group | Current/Former Smokers | Never Smokers
Number analyzed (Participants) | 26 | 23
participants
  Adverse Events | 26 | 23
  Serious Adverse Events | 14 | 7

ADVERSE EVENTS:
Time Frame: Up to 2 Years
Arm/Group | Current/Former Smokers | Never Smokers
Serious Adverse Events (participants affected / at risk) | 14/26 | 7/23
Other Adverse Events (participants affected / at risk) | 26/26 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Current/Former Smokers (N=26) | Never Smokers (N=23)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Biopsy muscle (Investigations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Current/Former Smokers (N=26) | Never Smokers (N=23)
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Conjunctivitis (Eye disorders) | 2 | 0
Dry Eye (Eye disorders) | 2 | 2
Growth of eyelashes (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 14 | 11
Dysphagia (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 10 | 11
Vomiting (Gastrointestinal disorders) | 5 | 4
Asthenia (General disorders) | 8 | 8
Chest pain (General disorders) | 5 | 3
Fatigue (General disorders) | 4 | 4
Mucosal inflammation (General disorders) | 3 | 3
Oedema (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 7 | 3
Xerosis (General disorders) | 2 | 3
Hepatobiliary disorders (Hepatobiliary disorders) | 2 | 0
Paronychia (Infections and infestations) | 2 | 3
Pneumonia (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Injury, poisoning and procedural complication (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 8 | 7
Anorexia (Metabolism and nutrition disorders) | 8 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Dysgeusia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 2 | 0
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 | 3
Dysuria (Renal and urinary disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 19 | 19
Skin fissures (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 2 | 1
Trichomegaly (Congenital, familial and genetic disorders) | 0 | 2
Blepharitis (Eye disorders) | 1 | 1
Mucosal dryness (General disorders) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 1
Surgical and medical procedures (Surgical and medical procedures) | 0 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 1

LIMITATIONS AND CAVEATS:
Treatment was ongoing for 3 patients at the time of the Clinical Study Report (CSR) cut-off. In the addendum to the CSR, there were no findings for these 3 patients that deviated from those observed in the original report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.